CLINICAL TRIAL: NCT05994976
Title: Collection of Samples From Subjects With Various Skin Conditions and Healthy Volunteers for Molecular Characterization of Inflammatory Skin Diseases
Brief Title: Collection of Samples From Subjects With Various Skin Conditions and Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: INNO-5034
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acne; Atopic Dermatitis; Chronic Hand Eczema; Hidradenitis Suppurativa; Plaque Psoriasis; Palmoplantar Pustulosis
MeSH Terms: conditions — Acne Vulgaris; Dermatitis, Atopic; Hidradenitis Suppurativa; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, stool, saliva, skin sample, lipid, sebum, microbiome, microorganism, hair, draining fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Healthy volunteers: Healthy adults
  Interventions: Procedure: Blood samples collection; Procedure: Oral samples collection; Procedure: Hair samples collection; Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping); Procedure: Skin surface material samples; Procedure: Drainage fluid samples collection; Procedure: Stool samples collection
- Acne: Adult subjects aged 18 to 45 years old with acne
  Interventions: Procedure: Blood samples collection; Procedure: Oral samples collection; Procedure: Hair samples collection; Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping); Procedure: Skin surface material samples; Procedure: Drainage fluid samples collection; Procedure: Stool samples collection
- AD: Adult subjects with Atopic Dermatitis (AD)
  Interventions: Procedure: Blood samples collection; Procedure: Oral samples collection; Procedure: Hair samples collection; Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping); Procedure: Skin surface material samples; Procedure: Drainage fluid samples collection; Procedure: Stool samples collection
- CHE: Adult subjects with Chronic Hand Eczema (CHE)
  Interventions: Procedure: Blood samples collection; Procedure: Oral samples collection; Procedure: Hair samples collection; Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping); Procedure: Skin surface material samples; Procedure: Drainage fluid samples collection; Procedure: Stool samples collection
- HS: Adult subjects with Hidradenitis suppurativa (HS)
  Interventions: Procedure: Blood samples collection; Procedure: Oral samples collection; Procedure: Hair samples collection; Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping); Procedure: Skin surface material samples; Procedure: Drainage fluid samples collection; Procedure: Stool samples collection
- PPP: Adult subjects with Palmoplantar pustulosis (PPP)
  Interventions: Procedure: Blood samples collection; Procedure: Oral samples collection; Procedure: Hair samples collection; Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping); Procedure: Skin surface material samples; Procedure: Drainage fluid samples collection; Procedure: Stool samples collection
- Psoriasis: Adult subjects with Psoriasis
  Interventions: Procedure: Blood samples collection; Procedure: Oral samples collection; Procedure: Hair samples collection; Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping); Procedure: Skin surface material samples; Procedure: Drainage fluid samples collection; Procedure: Stool samples collection

INTERVENTIONS:
Procedure: Blood samples collection — biomarkers and optional genetic analysis
Procedure: Oral samples collection — biomarkers analysis
Procedure: Hair samples collection — biomarkers analysis
Procedure: Skin samples collection (skin tape strip and/or skin biopsy, and/or skin scraping) — biomarkers analysis
Procedure: Skin surface material samples — biomarkers analysis
Procedure: Drainage fluid samples collection — biomarkers analysis
Procedure: Stool samples collection — biomarkers analysis

SUMMARY:
The purpose of the study is to collect different samples for molecular characterization of inflammatory skin diseases.

DETAILED DESCRIPTION:
This study is being conducted to collect samples from subjects with various skin conditions as well as healthy volunteers. Collected samples may be used for different analyses including, but not limited to, biomarker and gene expression analyses.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Subject is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
2. Subject must be willing to comply with all study procedures and must be available for the duration of the study.

   Healthy volunteers:
3. Male or female subject aged 18 years or older, at the time of consent.
4. Subject is in good general health, according to the investigator's judgment.

   Subjects with Acne:
5. Male or female subject aged 18 to 45 years old, inclusive, at the time of consent.

   Subjects with AD:
6. Male or female subject aged 18 years or older, at the time of consent.
7. Subject has clinically confirmed diagnosis of active AD, according to Hanifin and Rajka criteria.

   Subjects with CHE:
8. Male or female subject aged 18 years or older, at the time of consent.
9. Subject has at least a 6-month history of CHE before Screening (information obtained from medical chart or subject's physician, or directly from the subject).

   Subjects with HS:
10. Male or female subject aged 18 years or older, at the time of consent.
11. Subject has a clinically confirmed diagnosis of active HS with a disease duration of ≥ 6 months before screening as determined by the investigator through subject interview and/or review of the medical history.

    Subjects with PPP:
12. Male or female subject aged 18 years or older at the time of consent.
13. Subject has at least a 6-month history of PPP as defined by the presence of pustules on palms and/or soles, but without evidence of infection on palms and soles (information obtained from medical chart or subject's physician, or directly from the subject).

    Subjects with psoriasis:
14. Male or female subject aged 18 years or older, at the time of consent.

Exclusion Criteria:

All subjects:

1. Subject is a female who is pregnant or who is planning to become pregnant during the study.
2. Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 200 healthy volunteers and approximately 300 subjects with acne, atopic dermatitis (AD), chronic hand eczema (CHE), hidradenitis suppurativa (HS), palmoplantar pustulosis (PPP), and/or psoriasis will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Untargeted biomarker approach with gene expression profile of skin samples | Day 1
Exploratory biomarker and gene expression analyses. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No